CLINICAL TRIAL: NCT02925325
Title: Music Therapy for Major Depressive Disorder Residual Symptoms
Acronym: MTMDDRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Responsible Party: Principal Investigator, Jorge J. González Olvera, Dr., Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INPRF_MUS_THER_MDD
Record Dates: First submitted 2015-04-16; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Music therapy; Residual symptoms
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Therapy (Experimental): Music therapy 8 weekly sessions
  Interventions: Behavioral: Music therapy
- Usual Treatment (Active Comparator): It is the usual medical treatment.
  Interventions: Other: Usual Treatment

INTERVENTIONS:
Behavioral: Music therapy — Music therapy (MT) treatment focuses on the use of 2 techniques of intervention: receptive MT and active MT. The work of receptive application is described as the use of prerecorded music or executed by the music therapist with effect on the patient, without the latter's active involvement in the psychotherapeutic process of musical creation. While the active application, both the music therapist and patient are involved in musical creation, for example, the use of voice, body and musical instruments (Muñoz, 2008). Contemplate their psychotherapeutic possibilities in 3 different dimensions of patient: body, emotional and social work, as explained above. Treatment with MT, as in cognitive behavioral therapy, includes breathing exercises, stress-relaxation techniques, psychoeducation, and exercises for the management of irrational thoughts and erratic behavior patterns (Dobson and Dozois, 2010).
  Arms: Music Therapy
Other: Usual Treatment — It is the usual medical treatment that patients with major depressive disorder in remission but with residual symptom receives at the sponsor institution in a monthly basis.
  Arms: Usual Treatment

SUMMARY:
Residual Symptoms of Depression (SRD) are those symptoms that persist despite remission of MDD. They are characterized by a high incidence (approx. 90% of patients in remission) at the psychiatric clinic, have become a growing problem. Its presence is associated with a high probability of relapse / recurrence and disability, as determined by decreased performance and low quality of life. Their neglect has generated an increase in clinical and socioeconomic costs, alerting the need for research to provide treatment strategies. The application of different types of psychotherapy has been successful in abating SRD. The present study aims to evaluate the clinical changes related to the application of music therapy as a treatment of SRD, through a randomized controlled trial with two treatment arms trial. Music Therapy (MT) is a psychotherapy provided by specialized health professionals, and is defined as the clinical use of musical evidence-based interventions within a therapeutic relationship. MT treatment group will design an application schema of 8 sessions (2 hrs. Each) over a period of two months (one session per week). The control group will receive the Usual Treatment (TU) which corresponds to the usual clinical psychiatric treatment by the physician in the INPRF, with the same duration. The evaluation will be conducted with clinimetric testing at baseline, at the end of the track and after three months of treatment. This study seeks to identify the presence of SRD in a Mexican sample and explore a treatment designed for that purpose, also, show that the MT is a cost-effective implementation can become a new clinical option to extend the possibilities of assistance and deepen the investigation of this problem.

DETAILED DESCRIPTION:
GENERAL PURPOSE:

To evaluate the clinical changes related to the application of music therapy as a treatment for Residual Symptoms of Depression.

SPECIFIC OBJECTIVES:

1. Compare the pre and post treatment of residual symptoms by the HAM-D-21, BDI, SCL-90-R and CIDRS levels.
2. Compare the change of pre and post treatment obtained by the instruments for quality of life (WHOQOL-BREF), functioning (GAF and PSP) and perceived stress (PSS) values.

METHOD

Design - A randomized controlled trial with two treatment arms: the experimental group Music Therapy (MT); and control group Usual (TU) treatment. MT treatment group will design and will be completed in a period of two months, with an outline of 8 sessions (one per week). The TU corresponds to the usual clinical psychiatric treatment (drug) assigned by the attending physician in the INPRF.

POPULATION - patients attending the outpatient department of the National Institute of Psychiatry "Ramon de la Fuente" between 20 and 45, considered in remission of major depressive disorder (MDD) (DSM-IV) score ≤7 be included points on the Hamilton Depression Scale of (HAM-D-21) and / or ≤9 points in the Beck Depression Inventory (BDI), which have had a positive response to drug treatment and / or remain with pharmacotherapy phase continuation or maintenance, and there report or detection of persistent residual symptoms.

In this research, both participants in the control group and the experimental group, remain drug therapy throughout the study according to the instructions of the attending physician, so the period and type of administration shall be the sole decision of the same. In any case this protocol assessments will be conducted as planned. In the case of any change in drug therapy researchers take note of it for consideration in the final results.

SAMPLE SIZE - According to calculations made, the sample size is 48 patients. With an allocation of 24 patients in each treatment (MT and UT). It is considered to recruit an approximate previous historical studies in SRD sample (Fava et al., 1996; Fava et al., 1998).

To calculate the sample size formula for "comparison of two proportions" (Fernández, 2001), which was used as follows:

Where:

n = subjects required in each of the samples

Za = Z value corresponding to the desired risk

Zb = Z value corresponding to the desired risk

p1 = Value of the proportion in the control group, placebo control or usual treatment.

p2 = Value of the proportion in the group of the new treatment, intervention or technique.

p = average of the two proportions p1 and p2

The following data were considered:

* a confidence level of 95% or safety was established.
* A power of 80%.
* the effectiveness of standard treatment in preventing relapse (Fava et al was set at 32%., 1996; Paykel et al., 1999; Fava et al., 1998; Teasdale et al., 2000; Ma & Teasdale, 2004).
* was set at 70% of the desired effectiveness for MT in preventing relapse, considering the performance of psychotherapies reported (Fava et al., 1996; Paykel et al., 1999; Fava et al., 1998; Teasdale et al, 2000; Ma. & Teasdale, 2004).

This accounted for 15% of subjects the possible loss of the sample according to the following formula:

Losses set to n = (1/1-R) shows

n = number of subjects lossless

R = expected loss ratio

ELIGIBILITY:
Inclusion Criteria:

* Subsequent and file number at the National Institute of Psychiatry "Ramon de la Fuente" patients.
* Male or Female Patients.
* Age 20-45 years.
* Previous diagnosis of MDD according to DSM-IV.
* Presence of residual symptoms, with a score of ≤7 points in the HAM-D-21 and / or ≤9 points in BDI.
* Patients who agree to sign informed consent sheet.
* Patients without a psychotherapeutic treatment during the 8 weeks prior to baseline.
* Patients with any pharmacological antidepressant treatment in continuation phase or maintenance (Eg. SSRIs, benzodiazepines) with good adherence.

Exclusion Criteria:

* Patients with psychotic symptoms.
* Patients with suicidal risk.
* Patients with comorbid Axis I.
* Patients with comorbid Axis II as the primary diagnosis.
* Patients with any type of hearing chronic medical illness, neurological or (Eg. Hearing loss, tinnitus, etc.)
* Patients with addiction to any substance (except caffeine and nicotine).
* Patients with medical or psychological problems related to music (Eg. Amusia or musicogenic Epilepsy.
* Pregnant women.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 3 times: Baseline, Change from Baseline at the end of 2 Months Music Therapy and change from baseline at 3 months follow up
Clinical Interview for Depression and Related Syndromes | 3 times: Baseline, Change from Baseline at the end of 2 Months Music Therapy and change from baseline at 3 months follow up

SECONDARY OUTCOMES:
Symptom Checklist 90 Revised (SCL-90-R) | 3 times: Baseline, Change from Baseline at the end of 2 Months Music Therapy and change from baseline at 3 months follow up
Beck Depression Inventory | 3 times: Baseline, Change from Baseline at the end of 2 Months Music Therapy and change from baseline at 3 months follow up
WHO Quality of Life-BREF (WHOQOL-BREF) | 3 times: Baseline, Change from Baseline at the end of 2 Months Music Therapy and change from baseline at 3 months follow up
Personal and social performance scale (PSP) | 3 times: Baseline, Change from Baseline at the end of 2 Months Music Therapy and change from baseline at 3 months follow up
Perceived stress scale (PSS) | 3 times: Baseline, Change from Baseline at the end of 2 Months Music Therapy and change from baseline at 3 months follow up

OTHER OUTCOMES:
Global of Functioning Assessment Scale (GAF) | 3 times: Baseline, Change from Baseline at the end of 2 Months Music Therapy and change from baseline at 3 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Enrique O Flores Gutierrez, MD PhD, Study Chair — Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente; Jorge Julio González Olvera, MD PHD, Principal Investigator — Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Locations (1):
- Instituto Nacional de Psiquiatria Ramon de la Fuente Muñiz, Mexico City, Mexico City, Mexico